CLINICAL TRIAL: NCT04975737
Title: Multicenter, Double-blind, Randomized, Placebo-controlled Study of the Safety and Efficacy of the Subunit Recombinant Tuberculosis Vaccine GamTBvac in Preventing the Development of Respiratory Tuberculosis Not Associated With HIV Infection in Volunteers Aged 18-45 Years
Brief Title: Study of the Safety and Efficacy of the Subunit Recombinant Tuberculosis Vaccine GamTBvac
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gamaleya Research Institute of Epidemiology and Microbiology, Health Ministry of the Russian Federation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 02-GamTBvac-2020
Record Dates: First submitted 2021-07-09; First posted 2021-07-23 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2022-11

CONDITIONS: Tuberculosis
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vaccine Group (Experimental): 3590 volunteers who will receive 1 dose (0.5 ml) of the vaccine GamTBvac administered twice with an 8-week interval between administrations.
  Interventions: Biological: GamTBvac
- Placebo group (Placebo Comparator): 3590 volunteers who will receive 1 dose (0.5 ml) of the placebo administered subcutaneously twice with an 8-week interval between administrations.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: GamTBvac — The subunit recombinant tuberculosis vaccine GamTBvac (lyophilisate for preparation of solution for subcutaneous administration, 5.35 mg / dose)
  Arms: Vaccine Group
Biological: Placebo — Placebo for subcutaneous administration
  Arms: Placebo group

SUMMARY:
This is a multicenter, double-blind, randomized (in 1:1 ratio) placebo-controlled study to assess the safety and protective efficacy of the subunit recombinant tuberculosis vaccine GamTBvac against the development of respiratory tuberculosis not associated with HIV infection in volunteers aged 18-45 years.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female volunteers aged 18-45 years (inclusive);
2. Volunteers from population groups with a high incidence of tuberculosis (more than 30 people per 100 thousand population);
3. Absence of active tuberculosis, confirmed by chest x-ray or computed tomography;
4. Body mass index 18.5 - 30 kg / m2 (inclusive) according to Quetelet's weight and height index;
5. Signed informed consent to participate in the study in accordance with the current legislation;
6. Previous bacille Calmette Guerin (BCG) vaccination according to medical history or confirmed by the presence of a scar;
7. Absence of markers of the immune response to mycobacterial proteins ESAT6 and CFP10, which characterize the probable contact with M. tuberculosis prior to the start of the study confirmed by the tuberculosis skin test;
8. Negative pregnancy test in female volunteers with preserved reproductive potential at screening and on the day of the first vaccination;
9. Consent of male and female participants with preserved reproductive potential to observe an adequate method of contraception (double barrier method: male or female condom and combined hormonal contraceptive (oral, vaginal and transdermal forms can be used) or using a condom or diaphragm with spermicide during the entire period of vaccination and 1 month after completion of vaccination Exception: surgically sterile (more than 6 months) or postmenopausal (more than 12 months);
10. Consent of male participants not to participate in sperm donation during the entire period of vaccination and 1 month after completion of vaccination.

Non-inclusion criteria:

1. Positive test results for HIV-1/2 antibodies, HBsAg or hepatitis C antibodies at screening;
2. History of extrapulmonary tuberculosis;
3. History of chronic non-infectious respiratory disease, including idiopathic pulmonary fibrosis (IPF), bronchial asthma, chronic obstructive pulmonary disease (COPD), or pulmonary hypertension.
4. Clinically significant ECG abnormalities at screening;
5. Aggravated allergic history (bronchial asthma, history of anaphylaxis reactions);
6. Hypersensitivity to any component of the study drug or placebo; a history of drug intolerance;
7. History or presence of any disease or drug intake that, in the opinion of the investigator, may interfere with the assessment of the safety or efficacy of the vaccine.
8. History or presence of any possible immunodeficiency state according to physical and laboratory examination;
9. History of autoimmune disease (including systemic lupus erythematosus, type 1 diabetes, etc.);
10. Regular intake (lasting more than 2 weeks) of immunosuppressants or other immunomodulatory drugs less than 6 months before the start of the study (except the inhaled or topical forms of corticosteroids);
11. The use of immunoglobulin or blood products within 3 months before the start of the study or their planned appointment during the study;
12. Intake of antibacterial drugs within 14 days before vaccination (oral) and within 28 days before vaccination (parenteral);
13. Pregnancy, lactation, refusal to use double barrier method of contraception, woman's participation in an egg donation program;
14. Inability of the volunteer to understand the objectives, goals, research design, inability to comply with the prescribed protocol and schedule of visits and procedures;
15. Participation in clinical trials of medicinal products less than 3 months before the start of this study, or planned participation in another clinical trial;
16. Previous receipt of the GamTBvac vaccine and / or participation in clinical trials of any experimental anti-tuberculosis vaccines;
17. Any vaccination or planned vaccination less than a month before the first vaccination in this study or within a month after each vaccination in this study.
18. Anamnestic information about alcoholism, drug addiction, drug abuse;
19. Positive result of urine analysis for narcotic and psychotropic drugs;
20. Positive test for ethanol (exhaled air or using saliva test strips).

Exclusion Criteria:

Participation of a volunteer in the study may be terminated for the following reasons:

1. Development of primary tuberculosis of the respiratory system;
2. The researcher decided that the volunteer should be excluded in the interests of the volunteer himself;
3. The volunteer has a serious adverse event related to the study vaccine;
4. Failure to comply with the rules of participation in the study;
5. The participant refuses to cooperate or is undisciplined;
6. The participant was included in violation of the inclusion / non-inclusion criteria of the protocol;
7. Development of any other significant adverse events;
8. Deterioration of the volunteer's health.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 7180 (Estimated)
Dates: Start 2022-01-20 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Preventive efficacy (Ep) | 24 months after vaccination
  Preventive efficacy calculated as Ep=(1-RR)∗100%, where RR is the relative risk of developing pulmonary tuberculosis in the vaccine group compared to placebo

CONTACTS AND LOCATIONS:
Locations (1):
- City hospital #40, Saint Petersburg, Russia

IPD SHARING:
Plan to Share IPD: Undecided